CLINICAL TRIAL: NCT04229290
Title: Switching Treatment-Experienced, Integrase Inhibitor-Naïve, Virally Suppressed HIV-1 Infected Adults From Ritonavir Boosted Protease Inhibitors to Dolutegravir: An Open-Label Randomized Controlled Trial
Brief Title: Second-line Switch to Dolutegravir Study
Acronym: 2SD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nairobi (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Loice Achieng, Principal Investigator, University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2SD
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: HIV-1-infection
Keywords: HIV; Second-line; Switch; Protease inhibitor; Dolutegravir; Treatment experienced; Non-inferiority
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Randomised controlled, open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dolutegravir (Experimental): Participants in this arm will have a switch from a protease inhibitor based second line regimen to Dolutegravir maintaining the same NRTI backbone
  Interventions: Drug: Dolutegravir
- Protease Inhibitor (Active Comparator): Participants in this arm will be maintained on their protease inhibitor based second line regimen
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Switch of virally suppressed participants to Dolutegravir
  Other Names: DTG

SUMMARY:
Kenya has the 4th largest HIV burden in the world with about 1.6 million people living with HIV. Of these, just over 1 million are on antiretroviral therapy (ART). Current national guidelines recommend a first line regimen composed of 2 nucleoside reverse transcriptase inhibitors (NRTI) plus an integrase strand transfer inhibitor (INSTI) or a non-nucleoside reverse transcriptase inhibitor(NNRTI). Second line regimens are composed of 2 NRTI plus a ritonavir boosted protease inhibitor(PIr). This is based on evidence showing good clinical outcomes on this regimen. PIr are associated with side effects including an increase in cardiovascular disease risk and, have significant drug to drug interactions that complicate management of other conditions such as tuberculosis. INSTIs have been shown in one study to be an alternative to PIr in second line regimens when combined with fully active NRTIs. It is not clear if this would still be the case if the activity of the NRTIs was not known. The investigators will evaluate the efficacy of switching from a PIr to a dolutegravir based second line ART regimen.

Hypothesis: switching virologically suppressed patients from a PIr based second line to a dolutegravir based second line is non-inferior to continuing on a PIr based second line.

Objectives: The primary objective will be to evaluate the non-inferiority of switching to a DTG containing regimen relative to maintaining a PI/r containing second-line regimen in virologically suppressed, INSTI-naive HIV-1 positive adults (≥ 18 years old) as determined by having HIV-1 RNA ≥ 50 copies/ml at week 48. Secondary objectives will be to assess the impact of such a switch on CD4 count, safety and tolerability.

Methods: Open-label, randomized, non-inferiority, multisite trial over 48 weeks, describing the efficacy and safety of switching from a second-line ARV regimen containing a ritonavir-boosted protease inhibitor (PI/r) plus 2 NRTIs to DTG plus 2 NRTIs in patients with virological suppression (HIV-1 RNA < 50 copies/ml) for at least 12 weeks and with no prior INSTI exposure. Adult participants will be randomized at baseline to remain on their pre-enrollment PI/r or switch to DTG. Participants will continue the NRTIs from their pre-enrollment regimen in both arms. A total of 766 participants(388 per arm) will be recruited from 4 sites in Kenya Conclusion: This study seeks to inform guidelines around the efficacy and safety of alternative second line regimens.

DETAILED DESCRIPTION:
Background and Purpose of Research:

Current Kenya National Antiretroviral(ARV) Guidelines recommend that after failing an NNRTI-based first-line regimen, patients should move to a ritonavir-boosted protease inhibitor (PI/r) + 2 nucleoside reverse transcript inhibitors second-line regimen. Several randomised trials support this sequencing, even without drug resistance testing results to guide the choice of second-line NRTIs. The Kenya guidelines have recommended PI/r-based second-line regimens for over a decade and essentially all second-line patients in Kenya are currently on PI/r-based regimens with approximately 75% of these patients currently virally suppressed.

The pill burden, long-term toxicities, tolerability challenges, drug-drug interactions and higher cost of PI/r containing regimens are considerable disadvantages of the current second-line regimens in Kenya and much of sub-Saharan Africa. In contexts with high Tuberculosis (TB) prevalence, the impact of potential drug-drug interactions is considerable, requiring either super boosting of the PI with ritonavir which is toxic and poorly tolerated and only found to result in adequate drug levels for LPV/r but not for ATV/r or DRV/r or, use of rifabutin which is not co-formulated with other anti-mycobacterial agents and leads to a high pill burden affecting adherence. The supply of rifabutin has been unreliable in Kenya.

No study has evaluated a switch strategy from PI/r to DTG for virally suppressed treatment experienced patients who have failed a prior first line regimen consisting of a NNRTI + NRTIs. If such a strategy is found to be non-inferior to the current standard of care it would have major implications for the current regimens distribution in Kenya and similar settings, allowing a transition of almost 75% of current second-line patients from PI/r-based to DTG-based second line with lower cost, improved tolerability, decreased risk of toxicity, reduced risk of drug-drug interactions, and lower pill burden.

Summary of Previous Studies

A recent study has shown that a second-line regimen of dolutegravir (DTG) + 2 NRTIs is superior to LPV/r + 2 NRTIs after failing a first line regimen of NNRTI + 2 NRTIs in the presence of a fully active NRTI in the second line (Aboud 2019). The study excluded patients who did not have a fully active NRTI for second line, so the results can only be directly applied to scenarios where one can reliably predict activity of the NRTIs after first-line failure or where DRT results are available.

The Kenya National ARV Guidelines also recommend that patients on an alternative first line regimen, either NNRTI based or PI/r based, with virologic suppression should be switched to DTG/TDF/3TC. The evidence for this strategy comes from two studies showing that switch of virally suppressed patients to DTG-based first line regimens was associated with non inferior viral suppression, improved patient satisfaction and improved lipid profiles

In the NEAT022 study, investigators enrolled older individuals or those with high cardiovascular disease risk with the goal of analysing efficacy and impact of a change from a boosted PI to dolutegravir. Participants had suppressed HIV RNA while taking a boosted PI and two NRTIs, with no documented NRTI resistance mutations or previous virologic failure. All participants were over the age of 50 or had Framingham estimated 10-year risk of cardiovascular events greater than 10%. 415 individuals were randomised to continue two NRTI's plus a boosted PI or switch to dolutegravir while maintaining the same NRTIs. After 48 weeks, 97.5% of individuals in the boosted PI arm maintained virologic suppression compared to 94.5% in the dolutegravir switch arm (a non-statistically significant difference). Notably, lipid parameters and cardiovascular risk improved significantly in the switch arm.

Hypothesis Switch of virologically suppressed, INSTI-naïve HIV-1 positive adults (≥ 18 years old) on PI/r-based second line ARV regimens is non-inferior to continuing the PI/r-based regimen, as determined by risk of developing virological failure by 48 weeks.

Primary Objective To evaluate the non-inferiority of switching to a DTG containing regimen relative to maintaining a PI/r containing second-line regimen in virologically suppressed, INSTI-naive HIV-1 positive adults (≥ 18 years old) as determined by having HIV-1 RNA ≥ 50 copies/ml at week 48.

Secondary Objectives To assess the impact of switching to DTG on development of virological failure at week 24 To assess the impact of switching to DTG on maintenance of virological suppression at weeks 24 and 48 To assess the impact of switching to DTG on change in CD4 count at weeks 24 and 48 To assess the impact of switching to DTG on change in cardiovascular risk as determined by change in lipid values (total cholesterol, LDL, HDL, triglycerides and TC:HDL ratio) at weeks 24 and 48 and change in fasting blood glucose at weeks 24 and 48 To investigate the impact of switching to DTG on change in anthropometric measurements (weight, body-mass index, waist-hip ratio, waist circumference) To investigate the impact of switching to DTG on safety and tolerability To investigate the impact of switching to DTG on patient satisfaction, as determined by the HIV Treatment Satisfaction Questionnaire To investigate if outcomes differ based on the PI/r used To investigate if outcomes differ based on the NRTI used (TDF, ABC, or AZT) To investigate if outcomes differ for patients who switch NRTIs for clinical reasons during the study relative to patients who do not switch NRTIs during the study To investigate if outcomes differ based on if the NRTIs were changed from first-line to second-line To describe the genotypic resistance patterns for participants meeting protocol-defined virological failure

Study Design This is an open-label, randomized, non-inferiority, multicenter trial over 48 weeks, describing the efficacy and safety of switching from a second-line ARV regimen containing a ritonavir-boosted protease inhibitor plus 2 NRTIs to DTG plus 2 NRTIs in patients having achieved virological suppression for at least 12 weeks and with no prior INSTI exposure. Participants will be randomized at baseline to remain on their pre-enrollment PI/r or switch to DTG. Participants will continue the NRTIs from their pre-enrollment regimen in both arms.

Research Procedures Study visits will take place at screening, baseline, and weeks 4, 12, 24, 36, and 48 (with a 4-week extension as required for confirming HIV-1 RNA levels within the FDA snapshot window).

HIV-1 RNA viral load will be performed at screening and weeks 4, 12, 24 and 48. If HIV-1 RNA is ≥ 50 copies/ml then a repeat test will be performed at least two weeks after the detectable result to confirm virological failure. A repeat HIV-1 RNA result of ≥ 50 copies/ml is confirmed protocol-defined virological failure (PDVF) and genotypic resistance testing will be performed.

Other routine study investigations will include CD4, complete blood count, serum Creatinine, Alanine aminotransferase, Aspartate aminotransferase, total cholesterol, HDL, LDL, triglycerides, HBsAg, serum glucose, patient satisfaction questionnaires (HIVTSQ), and urine pregnancy test in women of child-bearing potential. In extenuating circumstances, such as travel restrictions or facility closures due to risk of COVID-19 infection or other unanticipated events, telephone calls may be used to complete as much information as possible on the CRFs for the scheduled study visits, and arrangements ade for laboratory samples to be taken at or near the subject's home.

A participant is free to withdraw from the study at any time. In addition, the investigators may decide, for reasons of medical prudence, to stop study medications. These participants will be followed to 48 weeks.

If any participants experience PDVF (two consecutive HIV-1 RNA levels of 50 copies/ml or more taken at least 14 days apart), the study PI/co-PI must be informed immediately for management recommendations, which will include genotypic drug resistance testing. Participants will be asked to attend all study visits.

Study medication may also be discontinued in the following instances:

If the participant withdraws their consent If the participant requires a substitution of the PI/r or DTG due to drug-drug interactions or toxicity. Changes to the NRTIs are allowed if clinically indicated, and changes within the PI/r class (e.g. from LPV/r to ATV/r) are allowed if it is required because of national supply chain limitations. Dose adjustments required to manage drug-drug interactions are allowed, following the product monograph for the drug If the investigators consider in the interest of the subject (i.e. intercurrent illness, unacceptable toxicity) that it is best for them to stop study medication The subject fails to comply with the protocol requirements, including poor adherence, or fails to cooperate with investigators

A female subject receiving DTG who becomes pregnant during the study must immediately have their DTG withdrawn to eliminate further exposure to the embryo/foetus. Exceptions may be discussed with Ethics and ViiV in situations where the benefits of continuing the pregnant woman on DTG outweigh the potential risks.

To minimize risk to subjects, study staff, and other staff at the study sites, precautions will be taken to reduce the risk of COVID-19 transmission in-line with the Ministry of Health guidelines and guidance from the Ethical Review Committee.

Source and Dose of the Products

Participants will be randomized to continue their pre-enrollment PI/r or switch from PI/r to DTG while continuing the NRTIs from the pre-enrollment regimen. Changes to the NRTIs are allowed throughout the study period only for clinical indications. Changes within the PI/r class are allowed (e.g. from LPV/r to ATV/r) if required by limitations in the national supply chain.

ARVs will be provided to all participants through the Kenya national ARV supply change mechanism, which uses generic fixed-dose combinations when available. For participants who are randomized to switch from PI/r+ABC/3TC to DTG+ABC/3TC, ViiV will provide the single-tablet fixed-dose combination of DTG/ABC/3TC in the commercial form of Triumeq®.

Participants who are randomized to take DTG will take a 50 mg tablet once daily, either as a single tablet in combination with a separate fixed-dose combination tablet of NRTIs or as part of a fixed-dose combination of DTG 50 mg and the NRTIs, as available through the national supply change or by ViiV (in the case of DTG/ABC/3TC).

Participants will be dispensed a 4 week supply of ARVs at baseline, an 8 week supply at week 4, and a 12 week supply at weeks 12, 24 and 36.

Number and Type of Participants

The anticipated sample size is 766 participants (383 per study arm). The sample size calculation is based on the primary endpoint of HIV-1 RNA ≥ 50 copies/ml at week 48 using the FDA snapshot method for the Intent-to-Treat Exposed (ITT-E) population. The sample size calculation assumes that the true difference in efficacy between treatment arms is zero and that overall virological failure rate is 3% at week 48. A total of 766 participants (383 participants per study arm) is required to provide at least 90% power to demonstrate non-inferiority for the DTG arm, compared to the control arm, with a one-sided significance level of 2.5% and non-inferiority margin of 4%.

Study Location:

All study sites are in Kenya and include: Kenyatta National Hospital, Thika Level 5 Hospital, Kiambu Level 5 Hospital and Jaramogi Oginga Odinga Teaching and Referral Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to understand and comply with the protocol requirements, instructions and restrictions
* Able and willing to give informed consent
* Age 18 years or above
* Documented HIV-1 infection as confirmed by HIV-antibody testing as per the Kenya National Guidelines
* Has been receiving a second-line ARV regimen containing a PI/r (DRV/r, ATV/r or LPV/r) and 2 NRTIs for at least 24 weeks
* Documented HIV-1 RNA viral load < 50 copies/ml at least 12 weeks prior to enrollment and no viral rebound between the first viral load < 50 copies/ml and the screening viral load
* HIV-1 RNA viral load < 50 copies/ml at screening (within 28 days prior to enrollment)
* If female and of childbearing potential, is using effective contraception and is willing to continue using effective contraception throughout the study period (as defined in Appendix 5). Note: Non-childbearing potential is defined as either post-menopausal (12 months of spontaneous amenorrhoea and age of 45 years or above) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy

Exclusion Criteria:

* Any prior use of integrase inhibitor
* Documented HIV-2 infection
* Using any concomitant therapy disallowed as per the reference safety information and product labelling for the study drugs
* Has AST and/or ALT at least 5-times greater than the upper limit of normal in conjunction with hepatitis B virus infection (HBV) or hepatitis C virus infection (HCV). Note: patients can enter the study with chronic HBV or HCV if AST and ALT are less than 5-times greater than the upper limit of normal and, in the investigators opinion, their medical status will not interfere with assessments or completion of the study
* Is both HBsAg positive and has a CrCl below 50 ml/min (as estimated using the Cockcroft-Gault estimate for glomerular filtration rate)
* Advanced renal insufficiency requiring dialysis
* If female, currently pregnant or breastfeeding, or intending to become pregnant during the study period
* Documented opportunistic infection within 4 weeks prior to the study enrolment
* Investigator opinion that the patient should switch from PI/r to DTG immediately for clinical reasons (including Grade 3 or 4 lipid abnormalities at screening or enrollment)
* Any condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the study
* History or presence of allergy to the study drugs or their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Virologic failure | 48 weeks
  Proportion of participants with HIV-1 RNA ≥ 50 copies/ml at week 48 (by US Food and Drug Administration snapshot algorithm, modified to allow for changes in NRTIs for clinical reasons)

SECONDARY OUTCOMES:
Virologic failure | 24 weeks
  Proportion of participants with HIV-1 RNA ≥ 50 copies/ml at week 24
Treatment success | 24 and 48 weeks
  Proportion of participants able to maintain virological suppression (HIV-1 RNA < 50 copies/ml with no discontinuation of the study treatment)
CD4 count | 24 and 48 weeks
  Change in CD4 count from baseline
Weight | 24 and 48 weeks
  Change in body weight from baseline
Body mass index | 24 and 48 weeks
  Change in body mass index from baseline
Waist-hip ratio | 24 and 48 weeks
  Change in waist-hip ratio from baseline
Waist circumference | 24 and 48 weeks
  Change in waist circumference from baseline
Blood sugar | 24 and 48 weeks
  Change in blood sugar from baseline
Total cholesterol | 24 and 48 weeks
  Change in blood total cholesterol from baseline
Low density lipoprotein | 24 and 48 weeks
  Change in low density lipoprotein from baseline
Triglyceride | 24 and 48 weeks
  Change in triglyceride from baseline
Total cholesterol:HDL ratio | 24 and 48 weeks
  Change in total cholesterol:HDL ratio from baseline
Percentage of participants experiencing an adverse event | 24 and 48 weeks
  clinical and laboratory adverse events
Resistance | 48 weeks
  Genotypic resistance mutations for participants with protocol-defined virological failure
Patient satisfaction: HIV Treatment Satisfaction Questionnaire scores | Baseline, week 24 and week 48
  HIV Treatment Satisfaction Questionnaire scores. Scores range from 0-60 with higher scores reflecting greater satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Loice Achieng, MD, MSC, Principal Investigator — University of Nairobi
Locations (4):
- Kenya (4):
  - Kiambu Level 5 Hospital, Kiambu
  - Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu
  - Kenyatta National Hospital, Nairobi
  - Thika Level 5 Hospital, Thika

IPD SHARING:
Plan to Share IPD: Yes
We will share IPD that underlie the results reported after de-identification (text, tables, figures and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after article publication and for a period of 36 months
Access Criteria: Researchers that provide a methodologically sound proposal and whose proposal has been approved by an independent review committee

REFERENCES:
- [Derived] Ombajo LA, Penner J, Nkuranga J, Mecha J, Mburu M, Odhiambo C, Ndinya F, Aksam R, Njenga R, Wahome S, Muiruri P, Eshiwani S, Kimani M, Ngugi C, Pozniak A. Second-Line Switch to Dolutegravir for Treatment of HIV Infection. N Engl J Med. 2023 Jun 22;388(25):2349-2359. doi: 10.1056/NEJMoa2210005. PMID 37342923